CLINICAL TRIAL: NCT02252458
Title: Can Fentanyl Lead to Opioid-induced Hyperalgesia in Healthy Volunteers? A Prospective, Randomized, Double-blinded Crossover Study
Brief Title: Can Fentanyl Lead to Opioid-induced Hyperalgesia in Healthy Volunteers?
Acronym: FentaOIH-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2014-054
Record Dates: First submitted 2014-09-08; First posted 2014-09-30 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Opioid induced hyperalgesia; Fentanyl
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl high dose (Experimental): Fentanyl 10mcg/kg of bodyweight
  Interventions: Drug: Fentanyl
- Fentanyl low dose (Active Comparator): Fentanyl 1mcg/kg of bodyweight
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl

SUMMARY:
The purpose of this study is to examine whether two clinically sensible dose regimen of fentanyl (low dose vs. high dose) lead to different pain scores as measured by the nonverbal rating scale (NRS) in healthy volunteers at 4.5 to 6.5 hours after fentanyl application. Pain modalities tested will include transdermal electrical stimulation and cold pressor pain.

The investigators hypothesize that the high dose fentanyl group will have an increase of approximately 20% in the NRS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (ASA I-II) male volunteers
* Age > 18 years
* BMI 18 - 25 kg/m2

Exclusion Criteria:

* Volunteers unable to give written informed consent
* Known drug allergies or intolerance to fentanyl
* Known drug allergies or intolerance to morphine and other opiates
* Recreational drug addiction or abuse
* Opiate use in the last month
* Volunteers taking confounding medication (analgesics, antihistamines, calcium or potassium channel blockers) in the last month
* History of motion sickness, neuropathy, chronic pain, neuromuscular or psychiatric disease
* Patients with renal failure (clearance < 30 ml/min)
* obstructive sleep apnea syndrome (OSAS)
* Indication for Rapid Sequence Induction
* Patients not understanding German, French, Italian or English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
COMPOSITE of pain scores as measured by the nonverbal rating scale (NRS) at 15 minute intervals within the timeframe specified below. | 4.5 to 6.5h after begin of fentanyl infusion

SECONDARY OUTCOMES:
Pain as measured by the nonverbal rating scale | 0-2h after begin of fentanyl infusion at 15 min intervals
cold pressor pain | at -15min, 1h, 2h, 3h, 4h, 5h, 6h, 6h30min after begin of infusion
Lab values (B-endorphin, fentanyl plasma Levels, potentially Adrenocorticotropic hormone (ACTH) / cortisol) | -15min, -10min, -5 min, 0 min, 15 min, 30 min, 45min, 1h, 1h 30min, 2h, 4h 30min, 4h 35min, 4h 40min, 4h 45min, 5h, 5h 30min, 6h, 6h 30min after begin of infusion
pupillary dilation response | baseline and at 4.5h after begin of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, PD Dr., MD, Principal Investigator — University Hospital Basel, Dep. of Anesthesia
Locations (1):
- Department of Anesthesia, University of Basel Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Mauermann E, Blum CA, Lurati Buse G, Bandschapp O, Ruppen W. Time course of copeptin during a model of experimental pain and hyperalgesia: A randomised volunteer crossover trial. Eur J Anaesthesiol. 2017 May;34(5):306-314. doi: 10.1097/EJA.0000000000000592. PMID 28106611